CLINICAL TRIAL: NCT06120660
Title: Musical Intervention on Stress Effects in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oviedo (Other)
Collaborators: Sociedad Española de Enfermería Intensiva y Unidades Coronarias (Unknown)
Responsible Party: Principal Investigator, Alba Maestro Gonzalez, Principal Investigator, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022.537; Investiga SEEIUC 2023 (Other: SEEIUC)
Record Dates: First submitted 2023-10-14; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Critical Care; Respiration, Artificial; Sedation
Keywords: music therapy; anxiety; critical care; nursing; stress, psychological; respiration, artificial
MeSH Terms: conditions — Respiratory Aspiration; Anxiety Disorders; Stress, Psychological | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group (Experimental): Music
  Interventions: Other: Music Therapy
- Control Group (No Intervention)

INTERVENTIONS:
Other: Music Therapy — Music Therapy
  Arms: Case Group

SUMMARY:
Aim: To evaluate the effects of a musical intervention on serum cortisol, prolactin, interleukin-6 levels and physiological parameters in sedated patients undergoing invasive mechanical ventilation.

DETAILED DESCRIPTION:
Design, Setting and Study Subjects: A randomized clinical trial will be conducted in the ICU of a spanish tertiary hospital. The study subjects will be adults, intubated, subjected to invasive mechanical ventilation, arterial catheter undergoing invasive mechanical ventilation, carrying an arterial catheter, with an adequate level of sedation and who do not present pain during the intervention.

Variables: The main variable will be total serum cortisol, prolactin, interleukin-6 levels. Secondary variables: secondary variables will be those used to measure physiological parameters to assess the patient's hemodynamic status of the patient in relation to the intervention.

Data collection: There will be 2 groups: intervention and control. The sample will be randomized as patients are admitted. First, they will be receiving the corresponding daily care. The first group of patients will receive the corresponding daily care. The patients in the intervention group will start the music therapy session through headphones, the patients in the control group will remain relaxed without any interruption during this time. All the variables will be collected before starting the study, during the study and at the end of the study.

Data analysis: A descriptive analysis of each variable will be performed. Subsequently, a bivariate analysis, previously checking the normality and homoscedasticity of the data.and homoscedasticity of the data. If statistically significant, post-hoc tests will be performed using Dunn's test.Dunn's test. Statistical significance will be accepted when p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Admitted to the ICU for a minimum of 24 hours
* Intubated patients undergoing invasive mechanical ventilation
* Arterial catheter carriers / central venous catheter
* Sedation level: BIS: 40 - 60
* No pain at the time of and during the procedure, which will be measured by a score of 0 on ESCID scale
* Not having previously undergone any other musical intervention.

Exclusion Criteria:

* Severe neurological disease or injury (CNS pathologies such as encephalitis, diffuse axonal injury, etc.)
* Severe psychiatric illness
* Suspected or confirmed drug or alcohol overdose/intoxication/abstinence
* Hearing impairment
* Skull lesions that preclude the use of headphones
* Patients with limitation of therapeutic effort or death expected within 24 hours
* Brain death diagnosis
* Failure to obtain informed consent from the legal representative within 72 hours of presentation
* Refusal of the responsible physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
levels of serum cortisol | Only one intervention per person will be performed. Serum levels will be measured before and after the intervention. That is, at minute 0 and 60.
  µg/dL
levels of prolactin | Only one intervention per person will be performed. Serum levels will be measured before and after the intervention. That is, at minute 0 and 60.
  ng/mL
levels of interleukin 6 | Only one intervention per person will be performed. Serum levels will be measured before and after the intervention. That is, at minute 0 and 60.
  pg/mL

SECONDARY OUTCOMES:
Bispectral Index (BIS) | Only one intervention per person will be performed. This variable will be recorded during the intervention, every 10 minutes. That is, at minute , 10, 20, 30, 40, 50 and 60.
  From 0 to 100
Blood Pressure | Only one intervention per person will be performed. This variable will be recorded during the intervention, every 10 minutes. That is, at minute , 10, 20, 30, 40, 50 and 60.
  mmHg
Heart rate | Only one intervention per person will be performed. This variable will be recorded during the intervention, every 10 minutes. That is, at minute , 10, 20, 30, 40, 50 and 60.
  bpm
Respiratory rate | Only one intervention per person will be performed. This variable will be recorded during the intervention, every 10 minutes. That is, at minute , 10, 20, 30, 40, 50 and 60.
  breaths per minute
Oxygen Saturation | Only one intervention per person will be performed. This variable will be recorded during the intervention, every 10 minutes. That is, at minute , 10, 20, 30, 40, 50 and 60.

CONTACTS AND LOCATIONS:
Overall Officials: Alba Maestro-González, Ph.D., Principal Investigator — University of Oviedo
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No
the data are confidential due to the sensitivity of the data

REFERENCES:
- [Background] Erdogan Z, Atik D. Complementary Health Approaches Used in the Intensive Care Unit. Holist Nurs Pract. 2017 Sep/Oct;31(5):325-342. doi: 10.1097/HNP.0000000000000227. PMID 28786890
- [Background] Umbrello M, Sorrenti T, Mistraletti G, Formenti P, Chiumello D, Terzoni S. Music therapy reduces stress and anxiety in critically ill patients: a systematic review of randomized clinical trials. Minerva Anestesiol. 2019 Aug;85(8):886-898. doi: 10.23736/S0375-9393.19.13526-2. Epub 2019 Apr 3. PMID 30947484
- [Background] Thaut MH. Music as therapy in early history. Prog Brain Res. 2015;217:143-58. doi: 10.1016/bs.pbr.2014.11.025. Epub 2015 Jan 31. PMID 25725914
- [Background] Seyffert S, Moiz S, Coghlan M, Balozian P, Nasser J, Rached EA, Jamil Y, Naqvi K, Rawlings L, Perkins AJ, Gao S, Hunter JD 3rd, Khan S, Heiderscheit A, Chlan LL, Khan B. Decreasing delirium through music listening (DDM) in critically ill, mechanically ventilated older adults in the intensive care unit: a two-arm, parallel-group, randomized clinical trial. Trials. 2022 Jul 19;23(1):576. doi: 10.1186/s13063-022-06448-w. PMID 35854358
- [Background] Kakar E, Billar RJ, van Rosmalen J, Klimek M, Takkenberg JJM, Jeekel J. Music intervention to relieve anxiety and pain in adults undergoing cardiac surgery: a systematic review and meta-analysis. Open Heart. 2021 Jan;8(1):e001474. doi: 10.1136/openhrt-2020-001474. PMID 33495383
- [Background] Khan SH, Wang S, Harrawood A, Martinez S, Heiderscheit A, Chlan L, Perkins AJ, Tu W, Boustani M, Khan B. Decreasing Delirium through Music (DDM) in critically ill, mechanically ventilated patients in the intensive care unit: study protocol for a pilot randomized controlled trial. Trials. 2017 Nov 29;18(1):574. doi: 10.1186/s13063-017-2324-6. PMID 29187230
- [Background] Khan SH, Kitsis M, Golovyan D, Wang S, Chlan LL, Boustani M, Khan BA. Effects of music intervention on inflammatory markers in critically ill and post-operative patients: A systematic review of the literature. Heart Lung. 2018 Sep-Oct;47(5):489-496. doi: 10.1016/j.hrtlng.2018.05.015. Epub 2018 Jul 9. PMID 30001799
- [Background] Taets GGC, Jomar RT, Abreu AMM, Capella MAM. Effect of music therapy on stress in chemically dependent people: a quasi-experimental study. Rev Lat Am Enfermagem. 2019 Jan 17;27:e3115. doi: 10.1590/1518-8345.2456.3115. PMID 30698217